CLINICAL TRIAL: NCT04161430
Title: A Phase III, Multicenter, Randomized, Double-Blind, Double-Dummy, Active-Comparator, Placebo-Controlled Clinical Trial of DBPR108 Tablets for Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Efficacy and Safety of DBPR108 100 mg in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPC/DBPR108201903/PRO-III-1
Record Dates: First submitted 2019-10-29; First posted 2019-11-13 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DBPR108; Type 2 diabetes mellitus; DPP4 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — DBPR108; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DRBP108 (Experimental): Phase A (Weeks 1-24): DBPR108 100mg + placebo matching Sitagliptin 100 mg; Phase B (Weeks 25-52): DBPR108 100 mg
  Interventions: Drug: DBPR108; Placebo matching sitagliptin
- Sitagliptin (Active Comparator): Phase A (Weeks 1-24): Placebo matching DBPR108 100 mg + Sitagliptin 100 mg; Phase B (Weeks 25-52): DBPR108 100 mg
  Interventions: Drug: Placebo matching DBPR108; Sitagliptin; DBPR108
- Placebo (Placebo Comparator): Phase A (Weeks 1-24): Placebo matching DBPR108 100 mg + placebo matching Sitagliptin 100 mg; Phase B (Weeks 25-52): DBPR108 100 mg
  Interventions: Drug: Placebo matching DBPR108; Placebo matching sitagliptin; DBPR108

INTERVENTIONS:
Drug: DBPR108; Placebo matching sitagliptin — Phase A (Weeks 1-24): DBPR108 100 mg once daily under fasted conditions for 24 weeks; Placebo matching sitagliptin 100 mg once daily under fasted conditions for 24 weeks.
  Phase B (Weeks 25-52): Drug: DBPR108 100 mg once daily under fasted conditions for 28 weeks.
  Arms: DRBP108
Drug: Placebo matching DBPR108; Sitagliptin; DBPR108 — Phase A (Weeks 1-24): Placebo matching DBPR108 100mg once daily under fasted conditions for 24 weeks; Sitagliptin 100 mg once daily under fasted conditions for 24 weeks.
  Phase B (Weeks 25-52): Drug: DBPR108 100 mg once daily under fasted conditions for 28 weeks.
  Arms: Sitagliptin
Drug: Placebo matching DBPR108; Placebo matching sitagliptin; DBPR108 — Phase A (Weeks 1-24): Placebo matching DBPR108 100 mg once daily under fasted conditions for 24 weeks; Placebo matching sitagliptin 100 mg once daily under fasted conditions for 24 weeks.
  Phase B (Weeks 25-52): Drug: DBPR108 100 mg once daily under fasted conditions for 28 weeks.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of 100 mg DRBP108 tablets in the treatment of type 2 diabetes mellitus. A total of 750 subjects will be randomly allocated to three groups: DRBP108, active comparator and placebo comparator, in a 3:1:1 ratio. The purpose of this study is to evaluate whether 24 weeks of DRBP108 treatment will adequately reduce hemoglobin A1C levels in T2DM subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the World Health Organization(WHO) (1999) criteria for the diagnosis and classification criteria for type 2 diabetes;
* 18 ≤ age ≤ 75 years old, male or female;
* 19kg/m^2 ≤ Body Mass Index（BMI ）≤ 35kg/m^2;
* Subjects with type 2 diabetes mellitus who did not regularly take oral hypoglycemic drugs at least 8 weeks before screening (i.e., continuous medication for <1 week);
* 7.0% ≤ HbA1c ≤ 9.5%;
* Subjects voluntarily participate in the trial and sign the informed consent form;
* Subjects agree to use contraception from the signing of the informed consent form to the end of 1 month of the last medication.

Exclusion Criteria:

* FPG > 13.9 mmol/L;
* A history of severe hypoglycemia (that is, hypoglycemia with severe cognitive impairment and requiring other measures to help recover);
* A history of allergy to similar drugs (DPP-4 inhibitors) or those who have been judged by the investigator to be allergic to tested drugs;
* Uncured hyperthyroidism or other diseases may cause secondary blood sugar elevation;
* Continuous use of glucocorticoids within 4 weeks prior to screening or may uninterrupted use glucocorticoids ≥14 days during the trial (except for external use and inhalation)
* Subjects with chronic bowel disease associated with inflammatory bowel disease, partial intestinal obstruction, or obvious digestive and absorption disorders;
* Subjects with infectious diseases(all positive for HBsAg, HBeAg, HBcAb, or positive for hepatitis C antibody, or positive for anti-HIV antibody); Female subjects of childbearing age are positive in pregnancy test or are lactating;
* Subjects with a history of alcoholism or drug abuse;
* Subjects have the clinically significant unstable diseases;
* Not suitable for this clinical trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c (%) compared to placebo comparator at week 24 | Baseline, week 24
  Change reflects the experimental value (baseline subtract) minus the placebo comparator value (baseline subtract) at week 24. HbA1c represents the percentage of glycosylated hemoglobin.

SECONDARY OUTCOMES:
Change from baseline in HbA1c (%) compared to active comparator at week 24 | Baseline, week 24
  Change reflects the experimental value (baseline subtract) minus the active comparator value (baseline subtract) at week 24. HbA1c represents the percentage of glycosylated hemoglobin.
The percentage of subjects with HbA1c≤6.5% and HbA1c≤7% at week 24 | Week 24
  Clinical response will be assessed by the percentage of subjects with HbA1c≤6.5% and HbA1c≤7% at week 24.
Change from baseline in HbA1c (%) at week 12, week 40, week 52 | Baseline, week 12, week 40, week 52
  Change reflects the experimental value minus the baseline value at week 12, week 40, week 52. HbA1c represents the percentage of glycosylated hemoglobin.
The percentage of subjects with HbA1c≤6.5% and HbA1c≤7% at week 12, week 40, week 52 | Week 12, week 40, week 52
  Clinical response will be assessed by the percentage of subjects with HbA1c≤6.5% and HbA1c≤7% at week 12, week 40, week 52.
Change from baseline in fasting plasma glucose/2-hour postprandial plasma glucose/body weight at week 12,week 24 | Baseline, week 12, week 24
  Change reflects the experimental value minus the baseline value in the fasting plasma glucose/2-hour postprandial plasma glucose/body weight at week 12,week 24. Plasma glucose was measured on a fasting basis or 2 hours after a standard meal, and is expressed as mmol/L. Body weight is expressed as kg.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Lou, Study Director — Department of Medicine, CSPC Clinical Development Division
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - the No, 1 People's Hospital of Changsha, Changsha, Huan Province